CLINICAL TRIAL: NCT04933500
Title: Comparative Study Between Dural Puncture Epidural Technique and Conventional Epidural Technique During Elective Gynecological Vaginal Surgeries
Brief Title: Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Organization: Cairo University (Other)
Other Study IDs: AL-2021
Record Dates: First submitted 2021-06-16; First posted 2021-06-21 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Anesthetic Regional Techniques for Vaginal Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional epidural: epidural needle: Tuhoy needle 1.3mm (18 G) with 20G multi-orifice epidural catheter
- Dural puncture epidural: epidural needle;Tuhoy needle 1.3mm (18G)with 20G multi-orifice epidural catheter and 25G Whitacre spinal needle
  Interventions: Device: Whitacre spinal needle

INTERVENTIONS:
Device: Whitacre spinal needle — 25G Whitacre spinal needle
  Groups: Dural puncture epidural

SUMMARY:
Both techniques are efficacious for sacral anesthesia during vaginal surgeries. Dural puncture epidural technique allows partial confirmation of epidural catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

  --Age(25-55)years
* Height(150-170cm)

Exclusion Criteria:

* patient refusal
* severe mitral or aortic stenosis

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult female Egyptian patients
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Onset of bilateral sacral sensory loss | 4months
  sacral sensory loss is observed by needle brick

CONTACTS AND LOCATIONS:
Locations (1):
- Abdelrahman, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No